CLINICAL TRIAL: NCT00133770
Title: A Pilot Study of Efficacy and Safety of Continuous Intravenous Infusion of Pantoprazole in the Treatment of Severe Erosive Esophagitis
Brief Title: Intravenous (IV) Pantoprazole in Erosive Esophagitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Qiang Cai MD/PhD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 259-2004; 3001K-200042 (Other Grant/Funding Number: Wyeth)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Esophagitis
Keywords: IV pantoprazole; Esophagitis
MeSH Terms: conditions — Esophagitis | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV pantoprazole (Experimental): The continuous IV pantoprazole compared to the once a day IV pantoprazole for 72 hours in the treatment of severe erosive esophagitis
  Interventions: Drug: pantoprazole

INTERVENTIONS:
Drug: pantoprazole — The continuous IV pantoprazole compared to the once a day IV pantoprazole for 72 hours in the treatment of severe erosive esophagitis
  Other Names: Protonix

SUMMARY:
The aim of this study is to examine whether pantoprazole (Protonix) given through continuous intravenous infusion for 72 hours is superior to Protonix given through once a day IV injection in the treatment of erosive esophagitis.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a very common disease that affects 20-50% of adults in Western Countries. The disease can be divided into three clinical categories: nonerosive reflux disease (NERD), erosive reflux disease (ERD), and Barrett's esophagus.

Intravenous (IV) infusion produces a faster and steadier acid suppression than an oral regimen. Furthermore, some patients with severe erosive esophagitis cannot take pills by mouth and will benefit from an IV formulation. Recently, we observed healing of severe erosive esophagitis with continuous IV pantoprazole in several patients in 3 days. The safety of IV pantoprazole has been demonstrated in patients with GERD, with Zollinger-Ellison syndrome, or bleeding ulcer. This study is to define the safety and efficacy of continuous IV pantoprazole in the treatment of severe erosive esophagitis.

Comparison: The continuous IV pantoprazole compared to the once a day IV pantoprazole for 72 hours in the treatment of severe erosive esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be men or non-pregnant women (a documented negative pregnancy test at enrollment for females of child bearing age) at least 18 years of age
* Patients who present with a severe erosive esophagitis - confirmed by endoscopy (a baseline endoscopy within 24 hours of study enrollment) to be grade five or six, with or without stricture and/or ulcer
* Patients or their legally authorized representatives must be capable of understanding or giving signed and dated informed consent before the study
* Patients with a high probability for compliance and completion of the study

Exclusion Criteria:

* Patients with less than grade five esophagitis
* Patients with esophagitis other than reflux esophagitis, such as infectious esophagitis and esophageal cancer
* Patients who present with gastrointestinal bleeding, hematocrit decrease greater than 6 units or require more than 2 units transfusion at the presentation or during the time of the study
* Patients with severe comorbidities, such as liver diseases with asparate transaminase (AST) or alanine transaminase (ALT) greater than 3 times upper limit normal (ULN); alkaline phosphatase greater than 5 times the ULN; total bilirubin greater than 3.0 mg/dl; kidney diseases with serum creatinine greater than 2.0 mg/dl in men or 1.6 mg/dl in women; heart diseases; lung diseases; sepsis; and airway intubation.
* Patients with history of glaucoma in either eye; history of any intraocular eye surgery within preceding 3 months; history of, or presence of, signs of optic nerve swelling; history of acute change in vision; or vision loss in either eye.
* Patients with any malignancy (except skin cancer) which required therapy within the last 6 months
* Patients with history of allergy to any proton-pump inhibitor (PPI) including pantoprazole
* Patients with known human immunodeficiency virus infection
* Patients with organ transplantation
* Patients without the ability to comply with the study protocol and complete the study in the judgment of the investigator
* Patients with prior administration of any PPI (within 72 hours) or histamine-2 receptor antagonist (within previous 24 hours) of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-07; Primary Completion 2006-07 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
the percentage of patients healed from severe esophagitis with IV pantoprazole at 7 days | 7 days
  the percentage of patients healed from severe esophagitis with IV pantoprazole at 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Cai, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States